CLINICAL TRIAL: NCT00119028
Title: Expanding and Testing VA Collaborative Care Models for Depression
Acronym: ReTIDES
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was withdrawn prior to enrollment.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: MNT 03-215; Project #0024; PCC # 2004-121657
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Major Depression; Post-Traumatic Stress Disorder
Keywords: Quality Improvement; Cluster Randomized Trial; Care Model
MeSH Terms: conditions — Depressive Disorder, Major; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other): Non-experimental QI intervention - No comparator
  Interventions: Procedure: Depression Care Quality Improvement Implementation

INTERVENTIONS:
Procedure: Depression Care Quality Improvement Implementation — We will used a randomized design to evaluate long term (18-month) cost effectiveness of TIDES collaborative care in six intervention clinics with fully-implemented collaborative care compared to three matched and randomly-assigned usual care clinics. We used a non-randomized quasiexperimental design (untreated control group with pretest and posttest) to measure impacts on clinician performance, knowledge, and attitudes in 6 newly-implemented collaborative care intervention clinics compared to 6 matched usual care clinics

SUMMARY:
Based on the published evidence, collaborative care for depression is both necessary and sufficient for improving care and outcomes for depressed patients in primary care settings. The Translating Initiatives in Depression into Effective Solutions (TIDES) project, upon which ReTIDES is based, developed a VA-adapted version of collaborative care through input from veterans, clinicians, and managers. The initial TIDES project resulted in a clinically stable and effective model as tested in seven primary care practices in three VISNs. This positive result provided the basis for spreading and sustaining the TIDES model and initiating the study of national implementation strategies and issues.

DETAILED DESCRIPTION:
Background:

Based on the published evidence, collaborative care for depression is both necessary and sufficient for improving care and outcomes for depressed patients in primary care settings. The Translating Initiatives in Depression into Effective Solutions (TIDES) project, upon which ReTIDES is based, developed a VA-adapted version of collaborative care through input from veterans, clinicians, and managers. The initial TIDES project resulted in a clinically stable and effective model as tested in seven primary care practices in three VISNs. This positive result provided the basis for spreading and sustaining the TIDES model and initiating the study of national implementation strategies and issues.

Objectives:

The objective of this grant was to carry out preparatory steps toward national implementation, including developing and investigating TIDES sustainability and partnering and marketing strategies. The project supported VISNs as learning organizations in the area of depression care improvement, and ultimately aimed to support as many as 8% to 10% of veterans nationally in improving their health and quality of life. Preparatory steps included 1) development of easily disseminated tools, including CPRS decision support, panel monitoring, and care manager and team training materials, 2) national and local dissemination to support TIDES model sustainability and spread and 3) evaluation using tools that would assess not only the success of this project, but could be used for quality monitoring during roll-out.

Methods:

Tools: We used the Chronic Illness Care model and Evidence Based Quality Improvement methods to develop tools for disseminating TIDES to additional medical centers and practices in 3 TIDES VISNs and two medical centers (with 10 practices) in one additional VISN. These tools were then used for national implementation. Dissemination: We served as technical expert consultants by 1) carrying out national and regional training; 2) linking to national patient care services, employee education, and information technology methods and priorities; and 3) supporting evidence-based quality improvement in new sites.We organized these efforts through a national dissemination plan.

Evaluation: We developed and applied 1) formative evaluation tools; 2) fine-tuned performance measure tools based on electronic data, and applied in a non-randomized quasi-experimental design (untreated control group with pretest and posttest); 3) a web-based survey for primary care clinicians and 4) an innovative implementation cost assessment approach. We also used 5) qualitative information on the process of dissemination , including links to national resources and 6) a randomized design to evaluate long term (18-month) cost effectiveness of TIDES.

Status:

Completed.

ELIGIBILITY:
Inclusion Criteria:

- Primary care providers at each participating site.

Exclusion Criteria:

- All providers not located at participating sites.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-04; Primary Completion 2008-12 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Impact of the intervention on depression performance measure, and provider attitudes. Quality of life-patient satisfaction. | 9/30/08

SECONDARY OUTCOMES:
Cost-effectiveness, system costs, tool kit development | 9/30/08

CONTACTS AND LOCATIONS:
Overall Officials: Lisa V. Rubenstein, MD MSPH, Principal Investigator — VA Greater Los Angeles Health Care System
Locations (6):
- United States (6):
  - Long Beach, Long Beach, California
  - VA Medical Center, Shreveport, Louisiana
  - VA Medical Center, Minneapolis, Minnesota
  - St. Cloud VA Medical Center, Saint Cloud, Minnesota
  - VA Medical Center, Cincinnati, Cincinnati, Ohio
  - Michael E DeBakey VA Medical Center, Houston, Texas

REFERENCES:
- [Result] Rubenstein LV, Meredith LS, Parker LE, Gordon NP, Hickey SC, Oken C, Lee ML. Impacts of evidence-based quality improvement on depression in primary care: a randomized experiment. J Gen Intern Med. 2006 Oct;21(10):1027-35. doi: 10.1111/j.1525-1497.2006.00549.x. Epub 2006 Jul 7. PMID 16836631
- [Result] Sherman SE, Fotiades J, Rubenstein LV, Gilman SC, Vivell S, Chaney E, Yano EM, Felker B. Teaching systems-based practice to primary care physicians to foster routine implementation of evidence-based depression care. Acad Med. 2007 Feb;82(2):168-75. doi: 10.1097/ACM.0b013e31802d9165. PMID 17264696
- [Result] Fickel JJ, Parker LE, Yano EM, Kirchner JE. Primary care - mental health collaboration: an example of assessing usual practice and potential barriers. J Interprof Care. 2007 Mar;21(2):207-16. doi: 10.1080/13561820601132827. PMID 17365393
- [Result] Campbell DG, Felker BL, Liu CF, Yano EM, Kirchner JE, Chan D, Rubenstein LV, Chaney EF. Prevalence of depression-PTSD comorbidity: implications for clinical practice guidelines and primary care-based interventions. J Gen Intern Med. 2007 Jun;22(6):711-8. doi: 10.1007/s11606-006-0101-4. PMID 17503104
- [Result] Chaney E, Rabuck LG, Uman J, Mittman DC, Simons C, Simon BF, Ritchie M, Cody M, Rubenstein LV. Human subjects protection issues in QUERI implementation research: QUERI Series. Implement Sci. 2008 Feb 15;3:10. doi: 10.1186/1748-5908-3-10. PMID 18279507
- [Result] Liu CF, Rubenstein LV, Kirchner JE, Fortney JC, Perkins MW, Ober SK, Pyne JM, Chaney EF. Organizational cost of quality improvement for depression care. Health Serv Res. 2009 Feb;44(1):225-44. doi: 10.1111/j.1475-6773.2008.00911.x. PMID 19146566
- [Result] Liu CF, Bolkan C, Chan D, Yano EM, Rubenstein LV, Chaney EF. Dual use of VA and non-VA services among primary care patients with depression. J Gen Intern Med. 2009 Mar;24(3):305-11. doi: 10.1007/s11606-008-0867-7. Epub 2008 Dec 20. PMID 19101777
- [Result] Smith JL, Williams JW Jr, Owen RR, Rubenstein LV, Chaney E. Developing a national dissemination plan for collaborative care for depression: QUERI Series. Implement Sci. 2008 Dec 31;3:59. doi: 10.1186/1748-5908-3-59. PMID 19117524
- [Result] Fickel JJ, Yano EM, Parker LE, Rubenstein LV. Clinic-level process of care for depression in primary care settings. Adm Policy Ment Health. 2009 Mar;36(2):144-58. doi: 10.1007/s10488-009-0207-1. Epub 2009 Feb 5. PMID 19194795
- [Result] Luck J, Hagigi F, Parker LE, Yano EM, Rubenstein LV, Kirchner JE. A social marketing approach to implementing evidence-based practice in VHA QUERI: the TIDES depression collaborative care model. Implement Sci. 2009 Sep 28;4:64. doi: 10.1186/1748-5908-4-64. PMID 19785754
- [Result] Foy R, Hempel S, Rubenstein L, Suttorp M, Seelig M, Shanman R, Shekelle PG. Meta-analysis: effect of interactive communication between collaborating primary care physicians and specialists. Ann Intern Med. 2010 Feb 16;152(4):247-58. doi: 10.7326/0003-4819-152-4-201002160-00010. PMID 20157139
- [Result] Parker LE, Ritchie MJ, Kirchner JE, Owen RR. Balancing health care evidence and art to meet clinical needs: policymakers' perspectives. J Eval Clin Pract. 2009 Dec;15(6):970-5. doi: 10.1111/j.1365-2753.2009.01209.x. PMID 20367694
- [Result] Rubenstein LV, Chaney EF, Ober S, Felker B, Sherman SE, Lanto A, Vivell S. Using evidence-based quality improvement methods for translating depression collaborative care research into practice. Fam Syst Health. 2010 Jun;28(2):91-113. doi: 10.1037/a0020302. PMID 20695669